CLINICAL TRIAL: NCT02785770
Title: A Phase 1, Single-dose, Randomized, 4-treatment, 4-period Crossover, Placebo- And Positive-controlled, Double-blind (Open-label For Positive Control), Sponsor-open Study To Determine The Effect Of PF-04447943 On Qtc Interval In Healthy Adult Subjects
Brief Title: A Study To Evaluate The Effect Of PF-04447943 On Qtc Interval In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: B0401018
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-06

CONDITIONS: Healthy
MeSH Terms: interventions — 6-(4-methyl-1-(pyrimidin-2-ylmethyl)pyrrolidin-3-yl)-1-(tetrahydro-2H-pyran-4-yl)-1,5-dihydro-4H-pyrazolo(3,4-d)pyrimidin-4-one; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-04447943 low dose (Experimental): 25 mg of PF-04447943
  Interventions: Drug: PF-04447943
- PF-04447943 high dose (Experimental): 100 mg of PF-04447943
  Interventions: Drug: PF-04447943
- Placebo (Placebo Comparator): Matching placebo for PF-04447943
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): 400 mg of moxifloxacin
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: PF-04447943 — Single oral dose of PF-04447943 administered as an extemporaneously prepared solution
  Arms: PF-04447943 high dose; PF-04447943 low dose
Drug: Placebo — Single oral dose of matching placebo for PF-04447943 administered as an extemporaneously prepared solution
  Arms: Placebo
Drug: Moxifloxacin — Single oral dose of moxifloxacin administered as tablet
  Arms: Moxifloxacin

SUMMARY:
This is a study designed to ascertain the effect of PF-04447943 on QT interval in healthy adult subjects. This is conducted as part of standard drug development.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non childbearing potential and/or healthy male subjects, between the ages of 18 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* History of cerebrovascular accident, transient ischemic attack (TIA), or traumatic brain injury.
* History of seizures or history or physical examination findings (eg localizing signs on neurologic examination) suggestive of structural central nervous system (CNS) abnormalities which may place patient at increased risk of seizures.
* History of orthostatic blood pressure changes or clinically significant orthostatic symptoms.
* Self reported history or risk factors for QT prolongation or torsades de pointes (eg, organic heart disease, congestive heart failure, hypokalemia, hypomagnesaemia, congenital long QT syndrome, myocardial ischemia or infarction), congenital deafness, family history of sudden death, and family history of long QT syndrome.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2016-10-20 (Actual); Study Completion 2016-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0401018&StudyName=A+Phase+1%2C+Single-dose%2C+Randomized%2C+4-treatment%2C+4-period+Crossover%2C+Placebo-+And+Positive-controlled%2C+Double-blind+%28open-label+For+Positive+Control%29%2C+Sponsor-open+Study+To+Determine+The+Effect+Of+Pf-04447943+On+Qtc+Interval+In+Healthy+Adult+Subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Moxifloxacin, Placebo, PF-04447943 100 mg, PF-04447943 25 mg: Participants received a single oral dose of Moxifloxacin 400 milligram (mg) tablet on Day 1 in the first intervention period; followed by a single dose of oral solution of placebo matched to PF-04447943 on Day 1 in the second intervention period; then a single dose of oral solution of PF-04447943 100 mg on Day 1 in the third intervention period; and then a single dose of oral solution of PF-04447943 25 mg on Day 1 in the fourth intervention period. A washout period of at least 7 days was maintained between each intervention period. Participants were followed up to 28 days after last dose of study medication.
- PF-04447943 25 mg, Moxifloxacin, Placebo, PF-04447943 100 mg: Participants received a single dose of oral solution of PF-04447943 25 mg on Day 1 in the first intervention period; followed by a single oral dose of Moxifloxacin 400 mg tablet on Day 1 in the second intervention period; then a single dose of oral solution of placebo matched to PF-04447943 on Day 1 in the third intervention period; and then a single dose of oral solution of PF-04447943 100 mg on Day 1 in the fourth intervention period. A washout period of at least 7 days was maintained between each intervention period. Participants were followed up to 28 days after last dose of study medication.
- Placebo, PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin: Participants received a single dose of oral solution of placebo matched to PF-04447943 on Day 1 in the first intervention period; followed by a single dose of oral solution of PF-04447943 100 mg on Day 1 in the second intervention period; then a single dose of oral solution of PF-04447943 25 mg on Day 1 in the third intervention period; and then a single oral dose of Moxifloxacin 400 mg tablet on Day 1 in the fourth intervention period. A washout period of at least 7 days was maintained between each intervention period. Participants were followed up to 28 days after last dose of study medication.
- PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin, Placebo: Participants received a single dose of oral solution of PF-04447943 100 mg on Day 1 in the first intervention period; followed by a single dose of oral solution of PF-04447943 25 mg on Day 1 in the second intervention period; then a single oral dose of Moxifloxacin 400 mg tablet on Day 1 in the third intervention period; and then a single dose of oral solution of placebo matched to PF-04447943 on Day 1 in the fourth intervention period. A washout period of at least 7 days was maintained between each intervention period. Participants were followed up to 28 days after last dose of study medication.
Period: Intervention Period 1 (1 Day)
Arm/Group | Moxifloxacin, Placebo, PF-04447943 100 mg, PF-04447943 25 mg | PF-04447943 25 mg, Moxifloxacin, Placebo, PF-04447943 100 mg | Placebo, PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin | PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin, Placebo
Started | 11 | 11 | 11 | 11
Completed | 11 | 11 | 11 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | Moxifloxacin, Placebo, PF-04447943 100 mg, PF-04447943 25 mg | PF-04447943 25 mg, Moxifloxacin, Placebo, PF-04447943 100 mg | Placebo, PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin | PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin, Placebo
Started | 11 | 11 | 11 | 11
Completed | 11 | 11 | 11 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Intervention Period 2 (1 Day)
Arm/Group | Moxifloxacin, Placebo, PF-04447943 100 mg, PF-04447943 25 mg | PF-04447943 25 mg, Moxifloxacin, Placebo, PF-04447943 100 mg | Placebo, PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin | PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin, Placebo
Started | 11 | 11 | 11 | 11
Completed | 11 | 10 | 10 | 11
Not Completed | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Family related obligations | 0 | 0 | 1 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | Moxifloxacin, Placebo, PF-04447943 100 mg, PF-04447943 25 mg | PF-04447943 25 mg, Moxifloxacin, Placebo, PF-04447943 100 mg | Placebo, PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin | PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin, Placebo
Started | 11 | 10 | 10 | 11
Completed | 11 | 10 | 10 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Intervention Period 3 (1 Day)
Arm/Group | Moxifloxacin, Placebo, PF-04447943 100 mg, PF-04447943 25 mg | PF-04447943 25 mg, Moxifloxacin, Placebo, PF-04447943 100 mg | Placebo, PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin | PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin, Placebo
Started | 11 | 10 | 10 | 11
Completed | 11 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Washout Period 3 (7 Days)
Arm/Group | Moxifloxacin, Placebo, PF-04447943 100 mg, PF-04447943 25 mg | PF-04447943 25 mg, Moxifloxacin, Placebo, PF-04447943 100 mg | Placebo, PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin | PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin, Placebo
Started | 11 | 10 | 10 | 10
Completed | 11 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Intervention Period 4 (1 Day)
Arm/Group | Moxifloxacin, Placebo, PF-04447943 100 mg, PF-04447943 25 mg | PF-04447943 25 mg, Moxifloxacin, Placebo, PF-04447943 100 mg | Placebo, PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin | PF-04447943 100 mg, PF-04447943 25 mg, Moxifloxacin, Placebo
Started | 11 | 10 | 10 | 10
Completed | 11 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis set included all participants who were randomized in the study.
Groups:
- Overall Study: All participants who were randomized to receive Moxifloxacin first, placebo first, PF-04447943 100 mg first and PF-04447943 25 mg first in intervention period 1.
Arm/Group | Overall Study
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 43

OUTCOME MEASURES:

1. Secondary Outcome: Time-Matched Mean Difference in Corrected QT Interval Using Fridericia's Correction Method (QTcF) for Moxifloxacin and Placebo
Description: Least square mean of QTcF measure for each reporting arm has been reported in summary or descriptive statistics. Least square mean difference across Moxifloxacin and placebo is reported in statistical analysis.
Time Frame: 0.5, 1 , 2, 3, 4, 8, 12 and 24 hours post-dose
Population: ECG analysis population included all participants randomized and treated who had at least 1 post-dose ECG measurement in at least 1 period.
Measure: Least Squares Mean (Standard Error); unit: Msec
Groups:
- Moxifloxacin 400 mg: Participants received a single oral dose of Moxifloxacin 400 mg tablet on Day 1 in any of the 4 intervention periods. Participants were followed up to 28 days after last dose of study medication.
- Placebo: Participants received a single dose of oral solution of placebo matched to PF-04447943 on Day 1 in any of the 4 intervention periods. Participants were followed up to 28 days after last dose of study medication.
Arm/Group | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 41 | 42
Msec
  0.5 Hour | 405.34 (0.9765) | 404.38 (0.9653)
  1 Hour | 411.98 (0.9765) | 404.09 (0.9653)
  2 Hours | 413.85 (0.9765) | 402.52 (0.9653)
  3 Hours | 413.03 (0.9765) | 404.43 (0.9653)
  4 Hours | 413.69 (0.9765) | 404.73 (0.9653)
  8 Hours | 406.72 (0.9765) | 398.66 (0.9653)
  12 Hours | 407.52 (0.9765) | 401.99 (0.9653)
  24 Hours | 406.81 (0.9765) | 403.06 (0.9653)
Statistical Analysis 1: Comparison: Moxifloxacin 400 mg vs Placebo; Moxifloxacin 400 mg versus Placebo, 0.5 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.4540, Repeated Measures Model; LS mean difference = 0.96, 90% CI 2-sided [-1.15 to 3.07]
Statistical Analysis 2: Comparison: Moxifloxacin 400 mg vs Placebo; Moxifloxacin 400 mg versus Placebo, 1 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Repeated Measures Model; LS mean difference = 7.88, 90% CI 2-sided [5.77 to 9.99]
Statistical Analysis 3: Comparison: Moxifloxacin 400 mg vs Placebo; Moxifloxacin 400 mg versus Placebo, 2 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Repeated Measures Model; LS mean difference = 11.33, 90% CI 2-sided [9.22 to 13.44]
Statistical Analysis 4: Comparison: Moxifloxacin 400 mg vs Placebo; Moxifloxacin 400 mg versus Placebo, 3 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Repeated Measures Model; LS mean difference = 8.59, 90% CI 2-sided [6.48 to 10.70]
Statistical Analysis 5: Comparison: Moxifloxacin 400 mg vs Placebo; Moxifloxacin 400 mg versus Placebo, 4 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Repeated Measures Model; LS mean difference = 8.96, 90% CI 2-sided [6.85 to 11.07]
Statistical Analysis 6: Comparison: Moxifloxacin 400 mg vs Placebo; Moxifloxacin 400 mg versus Placebo, 8 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Repeated Measures Model; LS mean difference = 8.07, 90% CI 2-sided [5.96 to 10.18]
Statistical Analysis 7: Comparison: Moxifloxacin 400 mg vs Placebo; Moxifloxacin 400 mg versus Placebo, 12 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Repeated Measures Model; LS mean difference = 5.53, 90% CI 2-sided [3.42 to 7.64]
Statistical Analysis 8: Comparison: Moxifloxacin 400 mg vs Placebo; Moxifloxacin 400 mg versus Placebo, 24 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.0036, Repeated Measures Model; LS mean difference = 3.74, 90% CI 2-sided [1.64 to 5.85]

2. Primary Outcome: Time-Matched Mean Difference in Corrected QT Interval Using Fridericia's Correction Method (QTcF) for PF-04447943 and Placebo at 0.5 Hour Post-Dose
Description: Least square mean of QTcF measure for each reporting arm has been reported in summary or descriptive statistics. Least square mean difference across PF-04447943 25 mg and placebo; PF-04447943 100 mg and placebo is reported in statistical analysis.
Time Frame: 0.5 hour post-dose
Population: Electrocardiogram (ECG) analysis population included all participants randomized and treated who had at least 1 post-dose ECG measurement in at least 1 period.
Measure: Least Squares Mean (Standard Error); unit: Millisecond (Msec)
Groups:
- PF-04447943 25 mg: Participants received a single dose of oral solution of PF-04447943 25 mg on Day 1 in any of the 4 intervention periods. Participants were followed up to 28 days after last dose of study medication.
- PF-04447943 100 mg: Participants received a single dose of oral solution of PF-04447943 100 mg on Day 1 in any of the 4 intervention periods. Participants were followed up to 28 days after last dose of study medication.
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 42
Millisecond (Msec) | 404.09 (0.9544) | 408.92 (0.9659) | 404.38 (0.9653)
Statistical Analysis 1: Comparison: PF-04447943 25 mg vs Placebo; PF-04447943 25 mg versus Placebo: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.8195, Repeated Measures Model; Least Square (LS) Mean Difference = -0.29, 90% CI 2-sided [-2.38 to 1.80]
Statistical Analysis 2: Comparison: PF-04447943 100 mg vs Placebo; PF-04447943 100 mg versus Placebo: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.0004, Repeated Measures Model; LS Mean Difference = 4.54, 90% CI 2-sided [2.44 to 6.64]

3. Primary Outcome: Time-Matched Mean Difference in Corrected QT Interval Using Fridericia's Correction Method (QTcF) for PF-04447943 and Placebo at 1 Hour Post-Dose
Description: as for outcome 2
Time Frame: 1 hour post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Msec
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 42
Msec | 404.23 (0.9544) | 409.14 (0.965) | 404.09 (0.9653)
Statistical Analysis 1: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9146, Repeated Measures Model; LS mean difference = 0.14, 90% CI 2-sided [-1.95 to 2.22]
Statistical Analysis 2: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.0001, Repeated Measures Model; LS mean difference = 5.04, 90% CI 2-sided [2.95 to 7.14]

4. Primary Outcome: Time-Matched Mean Difference in Corrected QT Interval Using Fridericia's Correction Method (QTcF) for PF-04447943 and Placebo at 2 Hours Post-Dose
Description: as for outcome 2
Time Frame: 2 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Msec
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 42
Msec | 403.76 (0.9544) | 406.78 (0.9659) | 402.52 (0.9653)
Statistical Analysis 1: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3272, Repeated Measures Model; LS mean difference = 1.24, 90% CI 2-sided [-0.84 to 3.33]
Statistical Analysis 2: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0009, Repeated Measures Model; LS mean difference = 4.26, 90% CI 2-sided [2.16 to 6.36]

5. Primary Outcome: Time-Matched Mean Difference in Corrected QT Interval Using Fridericia's Correction Method (QTcF) for PF-04447943 and Placebo at 3 Hours Post-Dose
Description: as for outcome 2
Time Frame: 3 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Msec
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 42
Msec | 403.95 (0.9544) | 406.69 (0.9659) | 404.43 (0.9653)
Statistical Analysis 1: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7024, Repeated Measures Model; LS mean difference = -0.48, 90% CI 2-sided [-2.57 to 1.60]
Statistical Analysis 2: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0768, Repeated Measures Model; LS mean difference = 2.26, 90% CI 2-sided [0.16 to 4.36]

6. Primary Outcome: Time-Matched Mean Difference in Corrected QT Interval Using Fridericia's Correction Method (QTcF) for PF-04447943 and Placebo at 4 Hours Post-Dose
Description: as for outcome 2
Time Frame: 4 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Msec
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 42
Msec | 402.76 (0.9544) | 405.94 (0.9659) | 404.73 (0.9653)
Statistical Analysis 1: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1201, Repeated Measures Model; LS mean difference = -1.97, 90% CI 2-sided [-4.06 to 0.12]
Statistical Analysis 2: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.3424, Repeated Measures Model; LS mean difference = 1.21, 90% CI 2-sided [-0.89 to 3.31]

7. Primary Outcome: Time-Matched Mean Difference in Corrected QT Interval Using Fridericia's Correction Method (QTcF) for PF-04447943 and Placebo at 8 Hours Post-Dose
Description: as for outcome 2
Time Frame: 8 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Msec
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 42
Msec | 397.31 (0.9544) | 398.55 (0.9659) | 398.66 (0.9653)
Statistical Analysis 1: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2870, Repeated Measures Model; LS mean difference = -1.35, 90% CI 2-sided [-3.44 to 0.74]
Statistical Analysis 2: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.9334, Repeated Measures Model; LS mean difference = -0.11, 90% CI 2-sided [-2.21 to 1.99]

8. Primary Outcome: Time-Matched Mean Difference in Corrected QT Interval Using Fridericia's Correction Method (QTcF) for PF-04447943 and Placebo at 12 Hours Post-Dose
Description: as for outcome 2
Time Frame: 12 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Msec
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 42
Msec | 399.83 (0.9544) | 399.38 (0.9659) | 401.99 (0.9653)
Statistical Analysis 1: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0893, Repeated Measures Model; LS mean difference = -2.16, 90% CI 2-sided [-4.24 to -0.07]
Statistical Analysis 2: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0412, Repeated Measures Model; LS mean difference = -2.61, 90% CI 2-sided [-4.71 to -0.51]

9. Primary Outcome: Time-Matched Mean Difference in Corrected QT Interval Using Fridericia's Correction Method (QTcF) for PF-04447943 and Placebo at 24 Hours Post-Dose
Description: as for outcome 2
Time Frame: 24 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Msec
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 42
Msec | 401.72 (0.9544) | 400.28 (0.9659) | 403.06 (0.9653)
Statistical Analysis 1: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2892, Repeated Measures Model; LS mean difference = -1.34, 90% CI 2-sided [-3.43 to 0.74]
Statistical Analysis 2: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0294, Repeated Measures Model; LS mean difference = -2.78, 90% CI 2-sided [-4.88 to -0.68]

10. Secondary Outcome: Time-Matched Mean Difference in Heart Rate for PF-04447943 and Placebo
Description: Least square mean of heart rate measure for each reporting arm has been reported in summary or descriptive statistics. Least square mean difference across PF-04447943 25 mg and placebo; PF-04447943 100 mg and placebo is reported in statistical analysis.
Time Frame: 0.5, 1 , 2, 3, 4, 8, 12 and 24 hours post-dose
Population: ECG analysis population included all participants randomized and treated who had at least 1 post-dose ECG measurement in at least 1 period. This outcome measure was planned not to be analyzed for reporting group: Moxifloxacin 400 mg.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute (bpm)
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 42
Beats per minute (bpm)
  0.5 Hour | 60.72 (0.6831) | 63.91 (0.6911) | 59.44 (0.6910)
  1 Hour | 60.98 (0.6831) | 64.43 (0.6911) | 58.60 (0.6910)
  2 Hours | 58.55 (0.6831) | 61.73 (0.6911) | 57.64 (0.6910)
  3 Hours | 58.37 (0.6831) | 61.21 (0.6911) | 58.68 (0.6910)
  4 Hours | 58.73 (0.6831) | 60.74 (0.6911) | 58.24 (0.6910)
  8 Hours | 61.13 (0.6831) | 63.40 (0.6911) | 61.95 (0.6910)
  12 Hours | 66.22 (0.6831) | 66.60 (0.6911) | 66.95 (0.6910)
  24 Hours | 59.32 (0.6831) | 60.23 (0.6911) | 62.35 (0.6910)
Statistical Analysis 1: Comparison: PF-04447943 25 mg vs Placebo; PF-04447943 25 mg versus Placebo, 0.5 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.1600, Repeated Measures Model; LS mean difference = 1.28, 90% CI 2-sided [-0.22 to 2.78]
Statistical Analysis 2: Comparison: PF-04447943 25 mg vs Placebo; PF-04447943 25 mg versus Placebo, 1 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.0092, Repeated Measures Model; LS mean difference = 2.38, 90% CI 2-sided [0.88 to 3.87]
Statistical Analysis 3: Comparison: PF-04447943 25 mg vs Placebo; PF-04447943 25 mg versus Placebo, 2 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.3174, Repeated Measures Model; LS mean difference = 0.91, 90% CI 2-sided [-0.59 to 2.41]
Statistical Analysis 4: Comparison: PF-04447943 25 mg vs Placebo; PF-04447943 25 mg versus Placebo, 3 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.7344, Repeated Measures Model; LS mean difference = -0.31, 90% CI 2-sided [-1.81 to 1.19]
Statistical Analysis 5: Comparison: PF-04447943 25 mg vs Placebo; PF-04447943 25 mg versus Placebo, 4 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.5881, Repeated Measures Model; LS mean difference = 0.49, 90% CI 2-sided [-1.00 to 1.99]
Statistical Analysis 6: Comparison: PF-04447943 25 mg vs Placebo; PF-04447943 25 mg versus Placebo, 8 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.3680, Repeated Measures Model; LS mean difference = -0.82, 90% CI 2-sided [-2.32 to 0.68]
Statistical Analysis 7: Comparison: PF-04447943 25 mg vs Placebo; PF-04447943 25 mg versus Placebo, 12 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.4200, Repeated Measures Model; LS mean difference = -0.73, 90% CI 2-sided [-2.23 to 0.76]
Statistical Analysis 8: Comparison: PF-04447943 25 mg vs Placebo; PF-04447943 25 mg versus Placebo, 24 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.0009, Repeated Measures Model; LS mean difference = -3.03, 90% CI 2-sided [-4.53 to -1.53]
Statistical Analysis 9: Comparison: PF-04447943 100 mg vs Placebo; PF-04447943 100 mg versus Placebo, 0.5 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Repeated Measures Model; LS mean difference = 4.46, 90% CI 2-sided [2.96 to 5.97]
Statistical Analysis 10: Comparison: PF-04447943 100 mg vs Placebo; PF-04447943 100 mg versus Placebo, 1 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Repeated Measures Model; LS mean difference = 5.83, 90% CI 2-sided [4.32 to 7.33]
Statistical Analysis 11: Comparison: PF-04447943 100 mg vs Placebo; PF-04447943 100 mg versus Placebo, 2 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p < 0.0001, Repeated Measures Model; LS mean difference = 4.09, 90% CI 2-sided [2.58 to 5.59]
Statistical Analysis 12: Comparison: PF-04447943 100 mg vs Placebo; PF-04447943 100 mg versus Placebo, 3 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.0059, Repeated Measures Model; LS mean difference = 2.53, 90% CI 2-sided [1.02 to 4.03]
Statistical Analysis 13: Comparison: PF-04447943 100 mg vs Placebo; PF-04447943 100 mg versus Placebo, 4 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.0063, Repeated Measures Model; LS mean difference = 2.50, 90% CI 2-sided [1.00 to 4.01]
Statistical Analysis 14: Comparison: PF-04447943 100 mg vs Placebo; PF-04447943 100 mg versus Placebo, 8 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.1138, Repeated Measures Model; LS mean difference = 1.45, 90% CI 2-sided [-0.06 to 2.95]
Statistical Analysis 15: Comparison: PF-04447943 100 mg vs Placebo; PF-04447943 100 mg versus Placebo, 12 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.6976, Repeated Measures Model; LS mean difference = -0.36, 90% CI 2-sided [-1.86 to 1.15]
Statistical Analysis 16: Comparison: PF-04447943 100 mg vs Placebo; PF-04447943 100 mg versus Placebo, 24 Hour: P-value was derived from repeated measures model with sequence, period, time, treatment and time-by-treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.0208, Repeated Measures Model; LS mean difference = -2.12, 90% CI 2-sided [-3.62 to -0.61]

11. Secondary Outcome: Time-Matched Mean Difference in PR Interval for PF-04447943 and Placebo
Description: Least square mean of PR interval measure for each reporting arm has been reported in summary or descriptive statistics. Least square mean difference across PF-04447943 25 mg and placebo; PF-04447943 100 mg and placebo is reported in statistical analysis.
Time Frame: 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Msec
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 42
Msec
  0.5 Hour | 171.59 (0.9261) | 170.52 (0.9361) | 172.24 (0.9358)
  1 Hour | 171.15 (0.9261) | 169.28 (0.9361) | 172.09 (0.9358)
  2 Hours | 170.43 (0.9261) | 169.72 (0.9361) | 171.60 (0.9358)
  3 Hours | 169.86 (0.9261) | 169.34 (0.9361) | 170.85 (0.9358)
  4 Hours | 170.59 (0.9261) | 169.22 (0.9361) | 171.16 (0.9358)
  8 Hours | 164.86 (0.9261) | 165.25 (0.9361) | 167.31 (0.9358)
  12 Hours | 166.08 (0.9261) | 165.48 (0.9361) | 166.49 (0.9358)
  24 Hours | 172.09 (0.9261) | 169.50 (0.9361) | 171.57 (0.9358)
Statistical Analysis 1: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.5760, Repeated Measures Model; LS mean difference = -0.64, 90% CI 2-sided [-2.53 to 1.25]
Statistical Analysis 2: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; p = 0.4126, Repeated Measures Model; LS mean difference = -0.94, 90% CI 2-sided [-2.83 to 0.95]
Statistical Analysis 3: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p = 0.3085, Repeated Measures Model; LS mean difference = -1.17, 90% CI 2-sided [-3.06 to 0.72]
Statistical Analysis 4: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 4]; Test type: Superiority or Other; p = 0.3889, Repeated Measures Model; LS mean difference = -0.99, 90% CI 2-sided [-2.88 to 0.90]
Statistical Analysis 5: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority or Other; p = 0.6192, Repeated Measures Model; LS mean difference = -0.57, 90% CI 2-sided [-2.46 to 1.32]
Statistical Analysis 6: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority or Other; p = 0.0332, Repeated Measures Model; LS mean difference = -2.45, 90% CI 2-sided [-4.34 to -0.56]
Statistical Analysis 7: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority or Other; p = 0.7224, Repeated Measures Model; LS mean difference = -0.41, 90% CI 2-sided [-2.30 to 1.48]
Statistical Analysis 8: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 8]; Test type: Superiority or Other; p = 0.6507, Repeated Measures Model; LS mean difference = 0.52, 90% CI 2-sided [-1.37 to 2.41]
Statistical Analysis 9: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 9]; Test type: Superiority or Other; p = 0.1366, Repeated Measures Model; LS mean difference = -1.72, 90% CI 2-sided [-3.62 to 0.18]
Statistical Analysis 10: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 10]; Test type: Superiority or Other; p = 0.0153, Repeated Measures Model; LS mean difference = -2.81, 90% CI 2-sided [-4.71 to -0.91]
Statistical Analysis 11: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 11]; Test type: Superiority or Other; p = 0.1040, Repeated Measures Model; LS mean difference = -1.88, 90% CI 2-sided [-3.78 to 0.02]
Statistical Analysis 12: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 12]; Test type: Superiority or Other; p = 0.1924, Repeated Measures Model; LS mean difference = -1.51, 90% CI 2-sided [-3.41 to 0.40]
Statistical Analysis 13: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 13]; Test type: Superiority or Other; p = 0.0928, Repeated Measures Model; LS mean difference = -1.94, 90% CI 2-sided [-3.84 to -0.04]
Statistical Analysis 14: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 14]; Test type: Superiority or Other; p = 0.0745, Repeated Measures Model; LS mean difference = -2.06, 90% CI 2-sided [-3.96 to -0.16]
Statistical Analysis 15: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 15]; Test type: Superiority or Other; p = 0.3836, Repeated Measures Model; LS mean difference = -1.01, 90% CI 2-sided [-2.91 to 0.90]
Statistical Analysis 16: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 16]; Test type: Superiority or Other; p = 0.0734, Repeated Measures Model; LS mean difference = -2.07, 90% CI 2-sided [-3.97 to -0.17]

12. Secondary Outcome: Time-Matched Mean Difference in QRS Interval for PF-04447943 and Placebo
Description: Least square mean of QRS interval measure for each reporting arm has been reported in summary or descriptive statistics. Least square mean difference across PF-04447943 25 mg and placebo; PF-04447943 100 mg and placebo is reported in statistical analysis.
Time Frame: 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose
Population: ECG analysis population included all participants randomized and treated who had at least 1 post-dose ECG measurement in at least 1 period. The outcome measure was planned not to be analyzed for reporting group: Moxifloxacin 400 mg.
Measure: Least Squares Mean (Standard Error); unit: Msec
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 42
Msec
  0.5 Hour | 90.76 (0.5481) | 89.28 (0.5547) | 89.96 (0.5544)
  1 Hour | 90.51 (0.5481) | 89.18 (0.5547) | 90.37 (0.5544)
  2 Hours | 90.89 (0.5481) | 89.14 (0.5547) | 89.88 (0.5544)
  3 Hours | 89.36 (0.5481) | 89.31 (0.5547) | 89.39 (0.5544)
  4 Hours | 89.84 (0.5481) | 88.95 (0.5547) | 91.02 (0.5544)
  8 Hours | 89.14 (0.5481) | 88.22 (0.5547) | 88.94 (0.5544)
  12 Hours | 89.61 (0.5481) | 89.09 (0.5547) | 89.58 (0.5544)
  24 Hours | 89.31 (0.5481) | 88.61 (0.5547) | 89.23 (0.5544)
Statistical Analysis 1: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.2588, Repeated Measures Model; LS mean difference = 0.80, 90% CI 2-sided [-0.36 to 1.96]
Statistical Analysis 2: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; p = 0.8465, Repeated Measures Model; LS mean difference = 0.14, 90% CI 2-sided [-1.03 to 1.30]
Statistical Analysis 3: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p = 0.1502, Repeated Measures Model; LS mean difference = 1.02, 90% CI 2-sided [-0.15 to 2.18]
Statistical Analysis 4: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 4]; Test type: Superiority or Other; p = 0.9700, Repeated Measures Model; LS mean difference = -0.03, 90% CI 2-sided [-1.19 to 1.14]
Statistical Analysis 5: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority or Other; p = 0.0947, Repeated Measures Model; LS mean difference = -1.18, 90% CI 2-sided [-2.34 to -0.02]
Statistical Analysis 6: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority or Other; p = 0.7759, Repeated Measures Model; LS mean difference = 0.20, 90% CI 2-sided [-0.96 to 1.36]
Statistical Analysis 7: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority or Other; p = 0.9649, Repeated Measures Model; LS mean difference = 0.03, 90% CI 2-sided [-1.13 to 1.19]
Statistical Analysis 8: Comparison: PF-04447943 25 mg vs Placebo; [analysis description as in outcome 10, analysis 8]; Test type: Superiority or Other; p = 0.9034, Repeated Measures Model; LS mean difference = 0.09, 90% CI 2-sided [-1.08 to 1.25]
Statistical Analysis 9: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 9]; Test type: Superiority or Other; p = 0.3391, Repeated Measures Model; LS mean difference = -0.68, 90% CI 2-sided [-1.85 to 0.49]
Statistical Analysis 10: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 10]; Test type: Superiority or Other; p = 0.0948, Repeated Measures Model; LS mean difference = -1.19, 90% CI 2-sided [-2.35 to -0.02]
Statistical Analysis 11: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 11]; Test type: Superiority or Other; p = 0.2959, Repeated Measures Model; LS mean difference = -0.74, 90% CI 2-sided [-1.91 to 0.43]
Statistical Analysis 12: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 12]; Test type: Superiority or Other; p = 0.9161, Repeated Measures Model; LS mean difference = -0.07, 90% CI 2-sided [-1.24 to 1.09]
Statistical Analysis 13: Comparison: PF-04447943 100 mg; [analysis description as in outcome 10, analysis 13]; Test type: Superiority or Other; p = 0.0036, Repeated Measures Model; LS mean difference = -2.07, 90% CI 2-sided [-3.24 to -0.91]
Statistical Analysis 14: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 14]; Test type: Superiority or Other; p = 0.3063, Repeated Measures Model; LS mean difference = -0.73, 90% CI 2-sided [-1.89 to 0.44]
Statistical Analysis 15: Comparison: PF-04447943 100 mg vs Placebo; [analysis description as in outcome 10, analysis 15]; Test type: Superiority or Other; p = 0.4918, Repeated Measures Model; LS mean difference = -0.49, 90% CI 2-sided [-1.65 to 0.68]
Statistical Analysis 16: Comparison: PF-04447943 100 mg; [analysis description as in outcome 10, analysis 16]; Test type: Superiority or Other; p = 0.3862, Repeated Measures Model; LS mean difference = -0.61, 90% CI 2-sided [-1.78 to 0.55]

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state.
Time Frame: Baseline (Pre-dose) up to 28 days after last dose of study drug (56 days)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 41 | 42
Participants
  AEs | 11 (27) [-0.36 to 1.96] | 9 [-1.85 to 0.49] | 8 | 8
  SAEs | 0 [-1.03 to 1.30] | 0 [-2.35 to -0.02] | 0 | 0

14. Secondary Outcome: Number of Participants With Physical Examination Abnormalities
Description: Full physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. Physical examination abnormalities were judged by the investigator.
Time Frame: Baseline (Pre-dose)
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 41 | 42
Participants | 1 (27) [-0.36 to 1.96] | 1 | 1 | 2

15. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Criteria for ECG abnormalities: maximum QTc corrected for heart rate using Bazett's formula (QTcB) and QTcF interval (450 to less than [<] 480 msec, 480 to <500 msec, greater than or equal to [>=] 500 msec; increase from baseline [IFB] >=30 msec and <60 msec, IFB >=60 msec). Baseline was defined as the average of the means obtained from the 3 sets of triplicate measurements taken at -1, -0.5 and 0 hours pre-dose on Day 1 within each intervention period.
Time Frame: Baseline up to 24 hours post-dose
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 41 | 42
Participants
  QTcB Interval 450 to <480 msec | 1 (27) [-0.36 to 1.96] | 3 [-1.85 to 0.49] | 1 | 0
  QTcB Interval 480 to <500 msec | 0 [-1.03 to 1.30] | 0 [-2.35 to -0.02] | 0 | 0
  QTcB Interval >=500 msec | 0 [-0.15 to 2.18] | 0 [-1.91 to 0.43] | 0 | 0
  QTcB IFB (>= 30 to <60) msec | 0 [-1.19 to 1.14] | 1 [-1.24 to 1.09] | 2 | 1
  QTcB IFB (>=60) msec | 0 [-2.34 to -0.02] | 0 [-3.24 to -0.91] | 0 | 0
  QTcF Interval 450 to <480 msec | 0 | 1 | 1 | 0
  QTcF Interval 480 to <500 msec | 0 | 0 | 0 | 0
  QTcF Interval >=500 msec | 0 | 0 | 0 | 0
  QTcF IFB (>=30 to <60) msec | 0 | 0 | 0 | 0
  QTcF IFB (>=60) msec | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Criteria for vital sign abnormalities: supine and standing pulse rate <40 bpm or greater than (>) 120 bpm, supine and standing systolic blood pressure (SBP) <90 millimeter of mercury (mmHg), supine and standing diastolic blood pressure (DBP) <50 mmHg, maximum (max.) increase from baseline (IFB) and decrease from baseline (DFB) in supine and standing SBP of >=30 mmHg, maximum IFB and DFB in supine and Standing DBP of >=20 mmHg.
Time Frame: Baseline (Pre-dose) up to 24 hours post-dose
Population: Safety analysis set included all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 41 | 42
Participants
  Supine SBP: <90 mmHg | 0 (27) [-0.36 to 1.96] | 0 [-1.85 to 0.49] | 0 | 0
  Standing SBP: <90 mmHg | 0 [-1.03 to 1.30] | 0 [-2.35 to -0.02] | 2 | 0
  Supine DBP: <50 mmHg | 0 [-0.15 to 2.18] | 0 [-1.91 to 0.43] | 1 | 0
  Standing DBP: <50 mmHg | 0 [-1.19 to 1.14] | 0 [-1.24 to 1.09] | 1 | 0
  Supine Pulse Rate: <40 bpm | 0 [-2.34 to -0.02] | 0 [-3.24 to -0.91] | 1 | 0
  Supine Pulse Rate: >120 bpm | 0 | 0 | 0 | 0
  Standing Pulse Rate: <40 bpm | 0 | 0 | 0 | 0
  Standing Pulse Rate: >120 bpm | 0 | 1 | 0 | 1
  Max. IFB in Supine SBP: >=30mmHg | 0 | 0 | 0 | 2
  Max. IFB in StandingSBP:>=30 mmHg | 1 | 0 | 0 | 1
  Max. IFB in Supine DBP: >=20 mmHg | 0 | 0 | 0 | 1
  Max. IFB in StandingDBP:>=20 mmHg | 2 | 2 | 3 | 1
  Max. DFB in Supine SBP:>=30 mmHg | 0 | 0 | 0 | 0
  Max. DFB in StandingSBP:>=30 mmHg | 2 | 1 | 1 | 3
  Max. DFB in Supine DBP:>=20 mmHg | 0 | 0 | 0 | 0
  Max. DFB in StandingDBP:>=20 mmHg | 2 | 4 | 1 | 0

17. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Hemoglobin(Hgb), hematocrit, red blood cell(RBC)<0.8*lower limit of normal(LLN), mean corpuscular(MC) Hgb, MC volume <0.9*LLN, >1.1*upper limit of normal(ULN), platelet<0.5*LLN,>1.75*ULN, lymphocyte, neutrophil<0.8*LLN, >1.2*ULN, basophil, eosinophil, monocyte>1.2*ULN, white blood cell(WBC)<0.6*LLN,>1.5*ULN, reticulocytes<0.5*LLN,>1.5*ULN; bilirubin>1.5*ULN, aspartate aminotransferase(AT), alanine AT, alkaline phosphatase>3.0*ULN, protein, albumin<0.8*LLN,>1.2*ULN; blood urea nitrogen, creatinine>1.3*ULN, uric acid>1.2*ULN; sodium<0.95*LLN,>1.05*ULN, potassium, chloride, calcium, bicarbonate<0.9*LLN,>1.1*ULN; glucose<0.6*LLN, >1.5*ULN, HbA1c>1.3*ULN, creatinine kinase>2*ULN; urine-specific gravity<1.003,>1.030, pH<4.5,>8, WBC, RBC>=20, bacteria>20, urobilinogen, glucose, ketone, protein, Hgb, nitrite, leukocyte esterase, bilirubin>=1; thyroid stimulating hormone<0.8*LLN,>1.2*ULN; cholesterol, triglycerides>1.3*ULN, high density lipoprotein cholesterol(DL-C) <0.8*LLN, low DL-C>1.2*ULN.
Time Frame: Baseline (Pre-dose) up to 24 hours post-dose
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Moxifloxacin 400 mg | Placebo
Number analyzed (Participants) | 43 | 42 | 41 | 42
Participants | 17 (27) [-0.36 to 1.96] | 12 [-1.85 to 0.49] | 12 | 18

18. Secondary Outcome: Maximum Plasma Concentration (Cmax) of PF-04447943
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose
Population: Pharmacokinetic (PK) parameter analysis population included all enrolled participants treated with PF-04447943 and who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg
Number analyzed (Participants) | 43 | 42
Nanogram per milliliter | 225.8 (19) [-0.36 to 1.96] | 947.3 (17) [-1.85 to 0.49]

19. Secondary Outcome: Time of Observed Maximum Plasma Concentration (Tmax) of PF-04447943
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose
Population: PK parameter analysis population included all enrolled participants treated with PF-04447943 and who had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: Hours
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg
Number analyzed (Participants) | 43 | 42
Hours | 1.0 (27) [0.500 to 3.0] | 1.02 [0.500 to 3.05]

20. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Time of Last Measurable Concentration (AUClast) of PF-04447943
Description: Area under the plasma concentration-time from time zero to time of last measurable concentration. Observed using the linear/log trapezoidal method.
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 3, 4, 8, 12 and 24 hours post-dose
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg
Number analyzed (Participants) | 43 | 42
Nanogram*hour per milliliter | 1454 (27) [-0.36 to 1.96] | 6277 (24) [-1.85 to 0.49]

ADVERSE EVENTS:
Time Frame: Baseline (Pre-dose) up to 28 days after last dose of study drug (56 days)
Description: Safety population included all participants who received at least 1 dose of study medication.
Arm/Group | PF-04447943 25 mg | PF-04447943 100 mg | Moxifloxacin 400 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42 | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 7/43 | 3/42 | 3/41 | 2/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04447943 25 mg (N=43) | PF-04447943 100 mg (N=42) | Moxifloxacin 400 mg (N=41) | Placebo (N=42)
Nausea (Gastrointestinal disorders) | 4 | 3 | 1 | 1
Headache (Nervous system disorders) | 3 | 2 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.